CLINICAL TRIAL: NCT04416529
Title: Tele-Mindfulness for Dementia's Family Caregivers: a Randomized Trial With a Usual Care Control Group
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 16-0216-E
Record Dates: First submitted 2020-05-25; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Caregivers; Mindfulness
Keywords: family caregivers; Dementia; mindfulness; Online; Internet-based
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: Participants were randomized to either the intervention group or the control group. All the participant were assessed at baseline, post-intervention and at 4-weeks follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (tele-MBCT) group (Experimental): Tele-MBCT was an 8-week program delivered to participants online via a videoconferencing program called Zoom by a tele-MBCT instructor. Tele-MBCT was delivered in three, 8-week rounds. Each round consisted of 8 weekly, 2-hour group sessions with 4-6 participants on Wednesdays from 2:00 to 4:00 pm. Participants were trained in mindfulness concepts and techniques including mindful eating, body scan, sitting meditation, breathing awareness, mindful walking and mindful movements. Participants were given a mindfulness a book called "The Mindful Way Workbook" and a practice log. The book was a guide for their daily practice at home and the practice log was a simple log for self-recording daily practices (number of minutes of daily MBCT practice) and a note pad for recording the reasons/obstacles for not practicing.
  Interventions: Behavioral: Tele-MBCT
- Control Group (No Intervention): Participants in the control group continued their usual caregiving activities.

INTERVENTIONS:
Behavioral: Tele-MBCT — Please see arm/group description.
  Arms: Intervention (tele-MBCT) group

SUMMARY:
Family caregivers were recruited through a combinations of strategies including a larger caregiving project and its partners, memory clinics, community outreach, online advertisement, flyers and brochures and word of mouth. After the telephone screening, eligible individuals were scheduled for an in-person baseline meeting at which they received additional information about the study, signed a consent form, completed baseline outcome measures and then were randomized to the intervention or control group using an online randomization program (http://www.graphpad.com/quickcalcs/index.cfm). All participants completed outcome measures immediately post-intervention for the intervention group and at 2 months for the control group and all participants completed follow-up outcome measures at 3 month following the baseline assessment. Participants in the intervention group completed a practice log which was designed to track their daily practice of mindfulness at home. The study was reviewed and approved by the Mount Sinai Hospital Research Ethics Board.

DETAILED DESCRIPTION:
Intervention (tele-MBCT) group Tele-MBCT was an 8-week program delivered to participants online via a videoconferencing program called Zoom. Zoom is an Ontario Personal Health Information Act (PHIPA) compliant videoconferencing program that provides remote communication for one-to-one or group meetings. Signing up, one-to-one meetings and attending a meeting as an invitee are free. The host of a group meeting is charged a monthly fee (CAD 14.99-19.99). All hosting fees were paid by the Sinai Health system.

Before starting the intervention, each participant's internet device was checked for compatibility with Zoom. If the device was not compatible, the participant was loaned a tablet for the duration of the intervention which was returned at the end of the study. Each participant was also trained in the use of their device to connect and use the Zoom platform and had an online intake interview with the tele-MBCT instructor.

Before each session, the host emailed the Zoom link to the participants. At the scheduled time of each group session, participants joined the live streamed session via their computers by using the link and following the on-screen instructions. During the live sessions, each participant was able to see, hear and speak with the group leader and other group members and they each could mute/unmute, turn on/off video, send messages via chat box and leave the session at any time if necessary.

The tele-MBCT instructor was a mental health clinician at the Reitman Centre who had a University of Toronto specialist and applied mindfulness certificate and mindfulness training at Mount Sinai Psychotherapy Institute (MSPI). She had extensive experience in developing and delivering online training and services to professionals and caregivers.

Participants in the intervention group were given a mindfulness package which included a book called "The Mindful Way Workbook" (Teasdale, Williams, and Segal 2014), a practice log and a snack pack of raisins (which was needed for the first session for mindful eating practice). "The Mindful Way Workbook" contains information about emotional distress, MBCT foundation and theories, other individuals' experiences with MBCT, weekly practices/explanations and homework. The book also contains a CD audio guide to each week's mindfulness practice. The practice log was a simple log for self-recording daily practices (number of minutes of daily MBCT practice) and a note pad for recording the reasons/obstacles for not practicing. These logs were anonymous and did not include any personal health information of the participants. At the completion of the tele-MBCT training, participants submitted their logs for analysis.

Tele-MBCT was delivered in three, 8-week rounds. Each round consisted of 8 weekly, 2-hour group sessions with 4-6 participants, held via Zoom on Wednesdays from 2:00 to 4:00 pm. For any technical problems during the sessions, participants had telephone access to the instructor.

During tele-MBCT training, participants were trained in mindfulness concepts and techniques including mindful eating, body scan, sitting meditation, breathing awareness, mindful walking and mindful movements. Mindfulness practices, except for mindful walking and mindful movements, were done in a sitting position in a chair or standing. Participants were asked to do the mindful walking with safety measures and in the room in which they were getting the training. The mindful movements were gentle stretches performed in seated and standing positions and were modified to each participant's abilities. At the completion of each session, participants were instructed to practice a specific mindfulness exercise during the week and record them in their practice log. They could use the CD for guided meditation and their home practice. The book also provided them with further readings. At the beginning of the training, participants were asked to set aside 30-45 minutes per day for practice. However, they were free to practice based on their schedule. Participants were permitted to miss up to 2 sessions for unanticipated problems. None of the sessions was audio/video recorded. Missed sessions were made up by reading about the missed session and doing the daily practice according to the book.

For this study, MBCT was modified in two ways for online delivery: omitting the retreat day from the schedule and mindful movements in lying position. In face to face MBCT training, the retreat day is held between sessions 6 and 7 and lasts 5-6 hours, during which individuals spend most of the day together in silence, doing guided practices of the previous sessions. Because of the long hours of the retreat day, it was deemed impractical in an online intervention and omitted. Because of safety issues, it was necessary that all the participants in the group could be seen (via their cameras) by the instructor during the whole training by adjusting the individual's device and finding the best position. This issue was addressed in the Zoom training and the interview with the instructor. Because doing the mindful movement in the lying position required adjustment of the device during the session which was time consuming and challenging, individuals were instructed to do mindful movements only in standing and sitting positions. However, the instructor explained the mindful movements in lying position and encouraged the participants to practice them at home.

Control Group Participants in the control group continued their usual caregiving activities. At 3 months after completion follow-up surveys, they received the "Mindful Way Workbook" and were offered the opportunity to attend the same tele-MBCT training after the study ended.

ELIGIBILITY:
Inclusion Criteria:

* Self-identification as a caregiver for a family member diagnosed with any type of dementia
* English literacy
* Access to a home computer connected to the Internet
* Basic familiarity with using a computer (the ability to check email and download files)
* Score at least 3 on the Single-item measure of self-perceived stress
* Agree to not engage in any formal community-based caregiver support programs, mind-body programs, or psychotherapy until they have completed training and follow-up evaluations

Exclusion Criteria:

* Active suicidality and self-harm ideas
* Recent diagnosis of major depression, severe anxiety, psychosis, and bipolar disorder
* Active substance misuse
* Starting on a new psychotropic medication within three months prior to entry into the study
* Involved in formal, professionally led meditation, yoga, or tai chi programs in the previous year

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-10-05 (Actual); Primary Completion 2017-09-07 (Actual); Study Completion 2017-11-07 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale (PSS)- 10-item version | Change from baseline at post-intervention for the intervention group and at 2 months for the control group and Change from baseline at 3 months for all participants
  Participant's level of stress

SECONDARY OUTCOMES:
Center for Epidemiologic Studies Depression Scale (CES-D) | Change from baseline at post-intervention for the intervention group and at 2 months for the control group and Change from baseline at 3 months for all participants
  Participant's symptoms of depression
State Anxiety Subscale of the Spielberger State-Trait Anxiety Inventory (STAI-S) | Change from baseline at post-intervention for the intervention group and at 2 months for the control group and Change from baseline at 3 months for all participants
  Current anxiety level
Coping Inventory for Stressful Situations- short form CISS-SF | Change from baseline at post-intervention for the intervention group and at 2 months for the control group and Change from baseline at 3 months for all participants
  Participants' coping responses to stressful situations
Self-compassion Scale (SCS) | Change from baseline at post-intervention for the intervention group and at 2 months for the control group and Change from baseline at 3 months for all participants
  Participants' level of self-compassion

OTHER OUTCOMES:
Demographics | At baseline
  Age, gender, level of education, employment status, marital status, care-recipient type of dementia, caregiver relationship, living status of the caregiver and care-recipient and length of time as a caregiver.
Feasibility criteria | Through study completion, an average of 1 year
  Recruitment, retention and compliance rates
Compliance rate | at 2 months (post-intervention) only for participants in the intervention group
  Participant compliance rates were evaluated based on attendance and practice rate, ability to complete the practice log and satisfaction questionnaire
Level of Satisfaction | at 2 months (post-intervention) only for participants in the intervention group
  Participants' level of satisfaction with the intervention based on the satisfaction questionnaire that was designed for this study

CONTACTS AND LOCATIONS:
Overall Officials: Joel Sadavoy, MD, FRCPC, Principal Investigator — Department of Psychiatry, University of Toronto

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zarei S, Lakhanpal G, Sadavoy J. Tele-Mindfulness for Dementia's Family Caregivers: A Randomized Trial with a Usual Care Control Group. Curr Alzheimer Res. 2022;19(5):364-372. doi: 10.2174/1567205019666220514131015. PMID 35570513